CLINICAL TRIAL: NCT03663725
Title: Phase III Randomised Trial Evaluating Treatment Intensification With Temozolomide in Adults With a Glioblastoma
Brief Title: Treatment Intensification With Temozolomide in Adults With a Glioblastoma
Acronym: StrateGlio
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Association de Neuro-Oncologues d'Expression Francaise (Other); Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: StrateGlio-1802; 2018-000410-38 (EudraCT Number)
Record Dates: First submitted 2018-09-04; First posted 2018-09-10 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma
Keywords: temozolomide; Stupp protocol
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensified protocol (Experimental): Early Temozolomide (TMZ) Concomitant TMZ Adjuvant TMZ Prolonged TMZ
  Interventions: Drug: Intensified protocol
- Stupp protocol (Active Comparator): Concomitant Temozolomide (TMZ) Adjuvant TMZ
  Interventions: Drug: Stupp protocol

INTERVENTIONS:
Drug: Intensified protocol — Early Temozolomide (TMZ) 1 cycle (150 mg/m²/ day X 5 days, per os) Started between day 2 and 15 after surgery/ biopsy RT (60 Gy, 2 Gy/fraction) + concomitant TMZ (75 mg/m2/day X 42 days, per os) Started between W4 and W6 after surgery/ biopsy Adjuvant TMZ 6 cycles (150-200 mg/m2 X 5 days /month, per os) Started 1 month after the end of the concomitant TMZ Prolonged TMZ Until progression, intolerance, patient's or physician's decision (150-200 mg/m2 every 4 weeks, per os)
  Arms: Intensified protocol
Drug: Stupp protocol — RT (60 Gy, 2 Gy/fraction) + concomitant Temozolomide (75 mg/m2/day X 42 days, per os) Started between W4 and W6 after surgery/ biopsy Adjuvant TMZ 6 cycles (150-200 mg/m2 X 5 days /month, per os) Started 1 month after the end of the concomitant TMZ
  Arms: Stupp protocol

SUMMARY:
Due to conflicting data on the optimal moment to start TMZ chemotherapy and the impact of prolongation of the adjuvant phase with TMZ, the ANOCEF (Association des Neuro-Oncologues d'Expression Francophone) group proposes this randomized trial comparing an intensified arm (early TMZ and extended adjuvant TMZ until toxicity, progression or patient refusal) versus the classical EORTC regimen as control (RT and concomitant TMZ started 4-6 weeks after surgery followed by a number of adjuvant TMZ cycles strictly limited to 6) for primary GBM adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18 years old
* Histological diagnosis of de novo GBM (extemporaneous diagnosis or standard pathological examination). In case of extemporaneous diagnosis, the patient can be included. If the diagnosis is not confirmed, the patient will be withdrawn from study.
* Time between initial surgery/biopsy and planned start of treatment (if allocated to the experimental arm) ≤ 15 days (ideally in the first 7 days)
* Karnofsky performance status (KPS) ≥ 60%, or KPS <60% only related to glioma-related motor paresis.
* Adequate biological functions
* Common toxicity criteria (CTC) non hematological adverse events ≤ Grade 1 (except for alopecia, nausea, vomiting and neurological symptoms)
* Females of child bearing potential must have a negative serum or urine pregnancy test within 7 days prior to initiation of treatment. Sexually active patients must agree to use adequate and appropriate contraception while on study drug and for 6 months after stopping the study drug.
* Standard radiation therapy deemed feasible (60 Gy, 30 fractions)
* Time interval of less than 43 days between initial surgery/biopsy and planned start of radiation therapy
* Written informed consent

Exclusion Criteria:

* Secondary or recurrent glioblastoma (GBM)
* Planned use of tumor-treating electric fields
* Planned use of Carmustine implants
* Prior malignancy in the last 5 years before inclusion or concomitant
* Severe myelosuppression
* Known hypersensitivity to any of the study drugs, study drug classes, excipients in the formulation or to dacarbazine (DTIC)
* Current or recent treatment with another experimental drug or patients included in a clinical therapeutic trial (in the 30 days prior to inclusion).
* Known current viral hepatitis, HIV infection or current active infectious disease
* Inability to swallow oral medications or any mal-absorption condition
* Pregnant or breastfeeding patients.
* Inability to comply with medical follow-up of the trial (geographical, social or psychic reasons)
* Person under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Estimated)
Dates: Start 2019-03-13 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | up to 18 months after recruitment of the last patient
  time interval from randomization to death whatever the cause

SECONDARY OUTCOMES:
Number of adverse events | up to 18 months after recruitment of the last patient
  from randomization until disease progression - reported and graded using the NCI-CTCAE v5.0 classification
Progression-free survival | up to 18 months after recruitment of the last patient
  time interval from randomization to the first occurrence of progression according to RANO criteria as assessed by the treating physician, or death whatever the cause

CONTACTS AND LOCATIONS:
Overall Officials: Florence LEFRANC, MD, Principal Investigator — ERASME; Bruno CHAUFFERT, MD, Principal Investigator — CHU Amiens
Locations (19):
- France (19):
  - Centre Hospitalier d'Amiens, Amiens
  - ICO Centre Paul Papin, Angers
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Hôpitaux Civils de Colmar, Colmar
  - Centre Georges François Leclerc, Dijon
  - CHU Grenoble Alpes, Grenoble
  - CHU de Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - CHU La Timone, Marseille
  - ICM Val d'Aurelle, Montpellier
  - CHRU Nancy, Nancy
  - ICO Centre René Gauducheau, Nantes
  - CHU de Nice - Hôpital de Cimiez, Nice
  - APHP La Pitié Salpêtrière, Paris
  - CH René Dubos, Pontoise
  - Institut Cancérologie Loire, Saint-Priest-en-Jarez
  - Centre Paul Strauss, Strasbourg
  - CHRU Tours, Tours

IPD SHARING:
Plan to Share IPD: No